CLINICAL TRIAL: NCT00607243
Title: Randomized, Double Blind, a Phase II/III Clinical Trial to Evaluate the Efficacy and Safety of CJ-50300 in Healthy Volunteers
Brief Title: Safety and Efficacy of CJ-50300 in Healthy Volunteers
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: HK inno.N Corporation (Industry)
Responsible Party: Principal Investigator, Myoung-don Oh, Professor, Division of Infectious Diseases, Department of Internal Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CJ_SPX_301; CJ corporation (Other: CJ corporation)
Record Dates: First submitted 2008-01-31; First posted 2008-02-05 (Estimated); Results first posted 2013-07-09 (Estimated); Last update posted 2013-07-09 (Estimated); Status verified 2013-07

CONDITIONS: Smallpox
Keywords: Smallpox vaccine efficacy
MeSH Terms: conditions — Smallpox

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional dose group (Experimental): Conventional CJ-50300 2.5 x 100000 pfu/dose vaccination
  Interventions: Biological: smallpox vaccine CJ-50300
- Low dose group (Experimental): Diluted CJ-50300 2.5 x 10000pfu/dose vaccination
  Interventions: Biological: smallpox vaccine CJ-50300

INTERVENTIONS:
Biological: smallpox vaccine CJ-50300 — Conventional dose group: 2.5 x 10 5 pfu/dose Diluted dose group:2.5 x 10 4 pfu/dose
  Other Names: CJ-53300

SUMMARY:
The currently available stock of smallpox vaccine would be insufficient in the face of an incident of smallpox attack. Thus, new manufacturing methods for smallpox vaccine are urgently needed because previous manufacturing methods using calf lymph are no longer acceptable in the view of current standards. Recently, CJ corporation in Republic of Korea has developed cell-culture derived smallpox vaccine (CJ-50300) which was manufactured by infecting MRC-5 cells. The aim of this clinical trial were to assess safety, reactogenicity, and immunogenicity of CJ-50300.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Korean male and female subjects between 20 and 60 years of age at the time of screening visit
2. Willing to participate and have signed the informed consent form
3. In good general health, without clinically skin diseases history, physical examination or laboratory test results
4. Hematocrit > 33% for women; > 38% for men
5. White cell count 3,300-12,000/mm3
6. Total lymphocyte count > 800 cells/mm3
7. Subjects who have never been vaccinated with smallpox vaccines

Exclusion Criteria:

1. Diseases or conditions that cause immunodeficiency (For examples; HIV AIDS, leukemia, lymphoma, generalized malignancy, agammaglobulinemia, history of transplantation, therapy with alkylating agents, antimetabolites, radiation, or oral or parenteral corticosteroids).
2. In close physical contact (household or at work) with an individual who has the diseases or conditions that cause immunodeficiency
3. History or present of eczema or atopic dermatitis
4. Allergy or sensitivity to any known components of vaccine or other medicines
5. In close physical contact (household or at work) with an individual who has acute or chronic skin conditions such as dermatitis, exfoliative dermatitis
6. Subjects requiring steroid therapy
7. Subjects who are taking immunosuppressive therapy
8. Subjects who are planning for blood donations
9. Autoimmune disease such as lupus erythematosus
10. Subjects who work in medical institution
11. Household contacts with women who are pregnant or breast-feeding
12. Female subjects who are pregnant or breast-feeding and have positive result by serum pregnancy test or urine pregnancy test, or do not using approved contraceptives such as sterilization, contraceptive ring injectable, combined oral contraceptive pills and barrier contraceptive, combined hormone-based therapy, contraceptive cream, contraceptive jelly, diaphragm or condoms
13. Subjects household member < 1 year old or work with children < 1 year old
14. Subjects with a known history of Cardiac disease or have three or more of the following risk factors: hyperpiesia, obesity, hyperlipidemia, glucosuria, sclerosis, cerebral arteriosclerosis
15. Receipt of immunoglobulin and steroid within 14 days of vaccination
16. Receipt of investigational research agents within 120 days of vaccination
17. HBsAg seropositive
18. HCV antibody seropositive
19. HIV seropositive
20. Subjects having fever (oral temperature > 38℃) or severe nutrition disorder
21. Blood donation within 12 weeks in advance screening visit
22. Subject who are not suitable to participate in study according to investigator's judgement

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Myoung-don Oh, M.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Jang HC, Kim CJ, Kim KH, Lee KH, Byun YH, Seong BL, Saletti G, Czerkinsky C, Park WB, Park SW, Kim HB, Kim NJ, Oh MD. A randomized, double-blind, controlled clinical trial to evaluate the efficacy and safety of CJ-50300, a newly developed cell culture-derived smallpox vaccine, in healthy volunteers. Vaccine. 2010 Aug 16;28(36):5845-9. doi: 10.1016/j.vaccine.2010.06.063. Epub 2010 Jun 30. PMID 20600480

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional-dose Group: Conventional CJ-50300 2.5 x 100000pfu/dose vaccination
- Low-dose Group: Diluted CJ-50300 2.5 x 10000pfu/dose vaccination
Period: Initial Post-vaccination Period
Arm/Group | Conventional-dose Group | Low-dose Group
Started | 82 | 41
Completed | 82 | 41
Not Completed | 0 | 0
Period: Telephone Safety Assessment Period
Arm/Group | Conventional-dose Group | Low-dose Group
Started | 82 | 41
Completed | 77 (80 Available for 3 months 77 Available for 6 months) | 39 (40 Available for 3 months 39 Available for 6 months)
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional-dose Group | Low-dose Group | Total
Number analyzed (Participants) | 82 | 41 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 82 | 41 | 123
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 23.9 (2.1) | 24.3 (2.8) | 24.0 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 61 | 28 | 89
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 82 | 41 | 123

OUTCOME MEASURES:

1. Primary Outcome: Cutaneous Take Reaction
Description: The "take reaction"was defined as a vesicular or pustular lesion or an area of definite palpable induration or congestion surrounding a central lesion (a crust or ulcer) occurring at the vaccination site at any of post-vaccination days (PVDs) 6-8. The vaccination site was photographed, and measures were taken.
Time Frame: 7-9 day
Measure: Number; unit: participants
Arm/Group | Conventional-dose Group | Low-dose Group
Number analyzed (Participants) | 82 | 41
participants | 81 [0.93 to 0.99] | 41 [0.90 to 1.00]

2. Primary Outcome: Adverse Reactions
Time Frame: 0-28 days
Reporting Status: Not Posted

3. Secondary Outcome: Antibody Response
Time Frame: 14 or 28 days
Reporting Status: Not Posted

4. Secondary Outcome: Cell-mediate Immunity
Time Frame: 14 or 28 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 28 days, 3 months, 6 months
Description: In the Conventional-dose Group, all 82 finished the 28 day follow up, 80 were available for 3 months, and 77 were available for the 6 months safety assessment.
  In the Low-dose Group, all 41 finished the 28 day follow up, 40 were available for 3 months, and 39 were available for the 6 months safety assessment.
Arm/Group | Conventional-dose Group | Low-dose Group
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/41
Other Adverse Events (participants affected / at risk) | 28/82 | 15/41
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Conventional-dose Group (N=82) | Low-dose Group (N=41)
Chill (Infections and infestations) | 8 | 5
Myalgia (Infections and infestations) | 7 | 8
Fatigue (Infections and infestations) | 16 | 9
Headache (Infections and infestations) | 9 | 8
Pain at vaccination site (Infections and infestations) | 17 | 10
Axillary pain or lymphadenopathy (Infections and infestations) | 28 | 15
Satellite lesion (Infections and infestations) | 8 | 4

LIMITATIONS AND CAVEATS:
the study was limited to vaccinia-naïve adults, thus yielding no data concerning the efﬁcacy of CJ-50300 in non-naïve adults or in children.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No